CLINICAL TRIAL: NCT02213952
Title: Efficacy of Autologous Platelet-Rich Plasma in the Treatment of Vascular Ulcers in Primary Care: Clinical Trial Phase III
Brief Title: PRP ULCERAS: Clinical Trial Phase III
Acronym: PRPULCERAS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Without recruitment
Sponsor: Basque Health Service (Other Government)
Collaborators: Osakidetza (Other)
Responsible Party: Principal Investigator, Kepa M. San Sebastián Moreno, Physician, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UIAPB-PRPULCERAS-2014-02; 2014-001514-26 (Other Grant/Funding Number: UIAPB-PRPULCERAS-2014)
Record Dates: First submitted 2014-07-16; First posted 2014-08-12 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Ulcer
Keywords: Ulcer; Platelet-Rich Plasma
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet-Rich Plasma (Experimental): Our goal is to evaluate the efficacy of the autologous Platelet-Rich Plasma (PRP) in the treatment of vascular ulcers, comparing to the conventional treatment (cure with humid environment), in primary care patients with chronic venous ulcer.
  Interventions: Drug: Platelet-Rich Plasma
- Usual treatment (Active Comparator): Usual treatment: Patients in the control group will be treated according to Osakidetza recommendations of humid environment cure. The choice of material for the cure depends on the prior assessment of the wound and surrounding skin, appearance and amount of exudate and the presence or absence of signs of infection. These cures will be performed every 48-72 hours.
  Interventions: Other: Usual treatment

INTERVENTIONS:
Drug: Platelet-Rich Plasma — For obtaining autologous PRP, will be drawn from 9-30 ml of blood of the patient in sterile tubes containing 4.5 ml of 3.8% sodium citrate. The tubes will be centrifuged for 8 min at 580 Gs to separate the different blood components according to density gradient. After centrifugation, we will aspire the PRP. We will add CaCl2 to the PRP (50l per ml of liquid plasma). While the plasma will get gelified, we will cure the ulcer with saline cleaning and mechanical removal. Then the ulcer will be covered with gelified PRP and a secondary dressing. This cure will be done each 7 days.
  Other Names: PRP
  Arms: Platelet-Rich Plasma
Other: Usual treatment — Usual treatment: Patients in the control group will be treated according to Osakidetza recommendations of humid environment cure. The choice of material for the cure depends on the prior assessment of the wound and surrounding skin, appearance and amount of exudate and the presence or absence of signs of infection. These cures will be performed every 48-72 hours.
  Other Names: Osakidetza protocol of humid environment cure.
  Arms: Usual treatment

SUMMARY:
INTRODUCTION: Vascular ulcers are an important pathology in the daily medical practice in all the assistance levels, and they have big repercussion referring to individual, social and labour levels, supposing a big consumption of human and material resources.The cure with autologous platelet rich plasma (autologous PRP) has demonstrated in different studies a decrease in the cicatrization time comparing to conventional methods in hospital levels, which becomes interesting contrasting its efficacy in primary care.

AIM:Evaluate the efficacy of the autologous PRP in the treatment of vascular ulcers, comparing to the conventional treatment ( cure with humid environment), in primary care patients with chronic venous insufficiency in C-6 degree (CEAP classification).

DESIGN: A study will be executed, which will consist in a randomized clinical test, multicentered, in parallel groups and opened. 150 patients suffering of venous vascular ulcers will be studied, who will be between the age of 40-100 years old, and who will be attached to 10 health centers. Variables for the identification, following, result and patient profile have been defined. Emphasize the variables of "ulcer area decreasing", "CIVIQ index", "% one cure per week".

DETAILED DESCRIPTION:
Vascular ulcers are an important pathology in the daily medical practice in all the assistance levels, and they have big repercussion referring to individual, social and labour levels, supposing a big consumption of human and material resources.The cure with autologous platelet rich plasma (autologous PRP) has demonstrated in different studies a decrease in the cicatrization time comparing to conventional methods in hospital levels, which becomes interesting contrasting its efficacy in primary care.The aim of this study is to evaluate the efficacy of the autologous PRP in the treatment of vascular ulcers, comparing to the conventional treatment (cure with humid environment), in primary care patients with chronic venous insufficiency in C-6 degree (CEAP classification). It is a study which will consist in a randomized clinical test, multicentered, in parallel groups and opened 150 patients suffering of venous vascular ulcers will be studied. Variables for the identification, following, result and patient profile have been defined. Emphasize the variables of "ulcer area change", "CIVIQ index", "% one cure per week".

ELIGIBILITY:
Inclusion Criteria:

* Patients from Barakaldo and Bilbao, who come to the treatment room at health centers in these towns belong to the OSI Ezkerraldea-Enkarterri-Cruces of Osakidetza-Basque Health Service.
* Men or women older than 18 years old.
* Patients with chronic venous insufficiency stage C-6 of the CEAP classification.
* Patients with vascular ulcers unresponsive to conventional treatment over a 2 months period or recurrence of previous venous ulcers.
* Patients who present an analytical before entering the studio, platelets and red blood cell count and hematocrit in normal range
* Ulcers whose diameter size is 30cm² or less.
* Greater Ankle Arm Index 0.8 and less than 1.5.
* Patients with recent analytic with number platelet and red blood cell count and hematocrit normal range.
* Patients with recent analytic negative to: Syphilis serology, Hepatitis B: HBsAg, Hepatitis C: Anti-HCV tests genomic nucleic acid amplification (NAT), HIV I / II: Anti-HIV I / II.
* Self or family support sufficient to move patients to the health center.
* Written informed consent of the patient

Exclusion Criteria:

* Patients on chronic immunosuppressive or retroviral.
* Coagulopathy
* Patients with chronic infectious diseases.
* Patients treated with radiotherapy or chemotherapy, or history of neoplasia.
* Patients with more than two active ulcers.
* Pregnant or childbearing potential not want to use contraception.
* Women breastfeeding.
* Patients with active infection or febrile syndrome at baseline.
* People who are taking a drug under clinical investigation or participated in any study under clinical investigation in the previous 30 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
ULCER SIZE CHANGE | Change from baseline at 9 weeks
  Change from baseline at 9 weeks of the surface area of the ulcer, in cm2, measured using ImageJ software from the weekly the photographs of the wound.

SECONDARY OUTCOMES:
QUALITY OF LIFE (INDEX CIVIQ) | Change from baseline at 9 weeks
  Change of the CIVIQ SCORE. 20-item self-reported quality of life questionnaire scale called Chronic Venous disease quality of life Questionnaire-20 (CIVIQ-20) was created and validated in France in 1996,1 as a sensitive instrument to capture the key dimensions of quality of life (QoL) specifically impaired by chronic venous disease (CVD). Four dimensions of the CIVIQ-20 were identified: physical (4 items), psychological (9 items), social (3 items), and pain (4 items).
Change of the percentage OF PATIENTS WITH A ONLY ONE TREATMENT FOR WEEK | Change from baseline at 9 weeks
  Change of the percentage OF PATIENTS WITH A ONLY ONE TREATMENT FOR WEEK

CONTACTS AND LOCATIONS:
Overall Officials: Kepa Mirena San Sebastian Moreno, Principal Investigator — C. Ezkerraldea Enkarterri.; Igone Hernández Cabezas., Study Chair — C. Ezkerraldea Enkarterri; Igone Lobato García, Study Chair — C. Ezkerraldea Enkarterri; Begoña Rodríguez Rodríguez., Study Chair — C. Bilbao; Ariadna Pérez Salvador, Study Chair — C. Ezkerraldea Enkarterri; Gonzalo Grandes Odriozola, Study Chair — Primary Care Research Unit of Bizkaia; Natalia Burgos Alonso., Study Director — Primary Care Research Unit of Bizkaia; Anna Giné March, Study Director — Primary Care Research Unit of Bizkaia; Kepa Mirena San Sebastian Moreno, Principal Investigator — C. Ezkerraldea Enkarterri
Locations (2):
- Spain (2):
  - Comarca Enkarterri Ezkerraldea, Portugalete, Bizakaia
  - UIAPB, Bilbao, Bizkaia

REFERENCES:
- [Derived] San Sebastian KM, Lobato I, Hernandez I, Burgos-Alonso N, Gomez-Fernandez MC, Lopez JL, Rodriguez B, March AG, Grandes G, Andia I. Efficacy and safety of autologous platelet rich plasma for the treatment of vascular ulcers in primary care: Phase III study. BMC Fam Pract. 2014 Dec 30;15:211. doi: 10.1186/s12875-014-0211-8. PMID 25547983